CLINICAL TRIAL: NCT00364910
Title: Post-Traumatic Stress Disorder (PTSD) Treatment in Cardiac Patients
Brief Title: Safety and Efficacy of Cognitive Behavior Therapy for People With Post-traumatic Stress and Cardiovascular Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 03-0985; R34MH071249 (NIH); 03-0985 DAHBR 96-BHC
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Myocardial Infarction (MI); Cognitive Behavioral Therapy (CBT); Adherence; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Myocardial Infarction; Depression | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral therapy (CBT) (Experimental): Participants will receive cognitive behavioral therapy
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)
- Educational session and treatment as usual (Active Comparator): Participants will receive an educational session and treatment as usual
  Interventions: Behavioral: Educational session and treatment as usual

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) — Participants meet with a therapist for three to five sessions brief exposure-based CBT.
  Arms: Cognitive behavioral therapy (CBT)
Behavioral: Educational session and treatment as usual — Participants assigned to the educational session attend one meeting with a researcher to discuss the results from their evaluation. They could also be referred to a mental health clinic of their choice to help relieve their symptoms.
  Arms: Educational session and treatment as usual

SUMMARY:
This study will evaluate the safety and efficacy of cognitive behavioral therapy in treating people who are experiencing post-traumatic stress disorder after a heart attack.

DETAILED DESCRIPTION:
PTSD usually develops in people who have experienced a traumatic or life-threatening event, including a health scare like a heart attack or catheterization. Symptoms of PTSD typically include anxiety, anger, and flashbacks or nightmares. PTSD symptoms are also associated with poor medical outcomes and nonadherence to medication after a heart attack. Fortunately, PTSD can sometimes be treated by antidepressants, anti-anxiety medication, and talk therapy. This study will compare the efficacy of cognitive-behavioral therapy (CBT) versus education and treatment as usual for treating people who are experiencing PTSD that is related to their cardiovascular illness (a heart attack or an invasive procedure such as catheterization).

Participants in this single-blind study will receive a psychiatric evaluation during which post-traumatic symptoms and feelings regarding their cardiovascular illness will be evaluated. Participants will then be randomly assigned to receive either CBT or a single educational session about PTSD, with up to 2 more follow-up educational meetings if needed. Participants assigned to the educational session will attend one meeting with a researcher to discuss the results from their evaluation. If they choose, they will also be referred to a mental health clinic for further care. Participants assigned to receive CBT will meet with a therapist once a week for at least 3 weeks. Participants will be offered the chance to meet with their therapist for two additional sessions if they need more time to discuss their symptoms. All participants will be re-evaluated at Months 2 and 6 using an interview, questionnaires,blood tests, blood pressure readings, and weight measurements.

ELIGIBILITY:
Inclusion Criteria:

* Suffered an acute heart attack or invasive treatment procedure related to a cardiovascular illness within 2 to 12 months of study entry
* Meets the threshold PTSD screening criterion
* Prescribed an anticoagulant or anti-aggregant at least 2 weeks prior to study entry

Exclusion Criteria:

* Readmitted to the hospital due to cardiovascular complications within 2 months of study entry
* Medically unstable
* Not prescribed aspirin
* Does not identify an event related to the cardiovascular illness as the primary trauma
* Cannot take care of self and is dependent on a caretaker for adherence to medications or clinic visits
* Suffers from other medical illnesses, including diseases that cause significant cognitive impairment (e.g., severe Alzheimer's), diseases that cause severe psychotic symptoms leading to disorientation (e.g., hepatic encephalopathy), diseases that cause brittle and uncontrollable blood pressure (e.g., pheochromocytoma), and diseases that cause uncontrollable hypercholesterolemia (e.g., severe familial hypercholesterolemia)
* Suicidal or history of suicide attempt
* Psychotic or suffers from a psychotic spectrum disorder
* Receiving psychotropic medications or psychotherapy and changed dosage or frequency of treatment within 2 weeks of study entry
* Currently receiving CBT

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Average blood pressure | Measured at Months 2 and 6
Impact of Event Scales (IES) | Measured at Months 2 and 6
  A 22-item self-report questionnaire measuring PTSD symptoms. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The IES-R yields a total score ranging from 0 (not at all) to 88 (extremely)

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | Measured at Months 2 and 6
  a 21 item self-report inventory measuring the severity of depression. Individuals are asked to respond to each question based on a two-week time period. Scoring is from 0 (minimal) to 3 (severe), with total score from 0-63. Higher total scores indicate more severe depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Shemesh, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Elmhurst Hospital Center, Queens, New York

REFERENCES:
- [Result] Shemesh E, Annunziato RA, Weatherley BD, Cotter G, Feaganes JR, Santra M, Yehuda R, Rubinstein D. A randomized controlled trial of the safety and promise of cognitive-behavioral therapy using imaginal exposure in patients with posttraumatic stress disorder resulting from cardiovascular illness. J Clin Psychiatry. 2011 Feb;72(2):168-74. doi: 10.4088/JCP.09m05116blu. Epub 2010 Apr 6. PMID 20441725